CLINICAL TRIAL: NCT03159585
Title: Application of NY-ESO-1-specific TCR Affinity Enhancing Specific T Cell Therapy (TAEST16001) in Solid Tumors Except Non Small Cell Lung Cancer,Including Liver Cancer,Gastric Cancer,Esophageal Cancer and so on.
Brief Title: To Evaluate the Efficacy of NY-ESO-1-specific T Cell Receptor Affinity Enhancing Specific T Cell in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Xiangxue Life Science Research Center (Unknown); Guangdong Xiangxue Precision Medical Technology Co., Ltd. (Industry); Xiangxue Pharmaceutical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-ZLZX-001
Record Dates: First submitted 2017-05-15; First posted 2017-05-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Liver Cancer Stage IV; Gastric Cancer Stage IV; Esophageal Cancer, Stage IV; Bone and Soft Tissue Tumors; Breast Cancer Stage IV; Bladder Carcinoma Stage IV; Prostate Carcinoma Stage IV; Thyroid Cancer Stage IV; Ovarian Cancer Stage IV; Solid Tumor
Keywords: TAEST16001
MeSH Terms: conditions — Liver Neoplasms; Stomach Neoplasms; Esophageal Neoplasms; Soft Tissue Neoplasms; Breast Neoplasms; Urinary Bladder Neoplasms; Prostatic Neoplasms; Thyroid Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: a single-center, open, single (or fractional) dose of safety and tolerability
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAEST16001 (Experimental): Patients who meet the inclusion criteria receive TAEST16001treatment after lymphodepleting by fludarabine and cyclophosphamide.
  Interventions: Drug: TAEST16001

INTERVENTIONS:
Drug: TAEST16001 — After completion of Lymphodepleting regimen pretreatment, the subject will receive an infusion of TAEST16001

SUMMARY:
The main purpose of this trial is to investigate the safety and tolerability of TAEST16001（TCR Affinity Enhancing Specific T cell Therapy）in the multi-line treatment failed advanced solid tumors except non small cell lung cancer,including liver cancer,gastric cancer,esophageal cancer,bone and soft tissue tumors,breast cancer, bladder carcinoma,prostate carcinoma,thyroid cancer, ovarian cancer and so on. The patients must meet the two criteria: human leukocyte antigens (HLA)-A*0201+ and NY-ESO-1 positive cells≥25% by immunohistochemistry.

DETAILED DESCRIPTION:
TCR-T cell therapy has made a breakthrough for tumors in recent years. Phase I/II trial of NY-ESO-1-specific TCR-T treatment for synovial sarcoma and melanoma, conducted by the Rosenberg team at the National Cancer Institute, showed that 61% Synovial cell sarcoma and 55% melanoma had benefits, without severe side effects found in T cell receptor (TCR) transduced T-Cell Immunotherapy. The US FDA has granted breakthrough TCR-T cell therapy for patients with inoperable or metastatic synovial sarcoma. The European Medicines Agency has also approved the same therapy to Priority Medicines(PRIME).

This clinical trial is mainly focused on cancer-testis antigen, because it is not expressed in normal cells. NY-ESO-1 antigen as one member of cancer-testis antigen, is commonly expressed in 10-50% of melanoma, lung, liver, esophageal, breast, prostate, bladder, thyroid and ovarian cancer cases, 60% of multiple myeloma cases, and 70-80% of synovial sarcoma. The NY-ESO-1 TCR cell therapy for synovial sarcoma and melanoma has benefited many patients, but its effect on other solid tumors is still unknown. So we plan to explore its efficacy in many types of solid tumors.

The trial is to investigate the safety and tolerability of TAEST16001 cell therapy in multi-line treatment failed advanced solid tumors except non small cell lung cancer,including liver cancer,gastric cancer,esophageal cancer,bone and soft tissue tumors,breast cancer, bladder carcinoma,prostate carcinoma,thyroid cancer, ovarian cancer and so on. The patients must meet the two criteria: HLA-A*0201+ and NY-ESO-1 positive cells≥25% by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* sign an informed consent before undertaking any trial-related activities;
* ≥18 and ≤75 years old;
* Multi-line treatment failed Solid Tumors except non small cell lung cancer,including Liver Cancer,Gastric Cancer,Esophageal Cancer,Bone and Soft Tissue Tumors,Breast Cancer, Bladder Carcinoma,Prostate Carcinoma,Thyroid Cancer, Ovarian Cancer and so on diagnosed by licensed pathologist;
* multi-line treatment failed patients;
* with measurable lesions according to Response Evaluation Criteria In Solid Tumors1.1 or immune related response criteria standard;
* meet the two screening indicators: HLA-A*0201+, NYESO-1+(≥25% by immunohistochemistry);
* Eastern Cooperative Oncology Group score 0-1;life expectancy is longer than 3 months;
* The patient did not receive anti-tumor therapy within 4 weeks before enrollment;
* A brain metastasis patient in a stable condition for one month after anti-tumor therapy can be included;
* left ventricular ejection fraction≥50%
* Lab test results meet the following requirements:

white blood cell count≥3.0×10^9/L; absolute neutrophil count≥1.5 ×10^9/L (No human granulocyte colony stimulating factor support); blood platelet≥75 ×10^9/L; Hemoglobin≥10g/dL (No transfusion in the last 7 days); Prothrombin time or International normalized rate ≤1.5×normal upper limit, except taking anticoagulant therapy; thrombin time≤1.5×normal upper limit, except taking anticoagulant therapy; a 24-hour creatinine clearance rate≥60mL/ min; Aspartate transaminase / serum glutamic oxaloacetic transaminase≤2.5 ×upper limit of normal; Alanine aminotransferase/ serum glutamate pyruvate transaminase≤2.5 ×upper limit of normal; total bilirubin≤1.5×upper limit of normal (expect that the subject has Gilbert's syndrome).

* no pregnant women；female patients must use contraceptive measures during the study and prohibit any homosexual or heterosexual;
* The patients can regularly visit the research institutions for related tests, evaluations, and management during the study period.

Exclusion Criteria:

* lung cancer ;
* received major surgery, conventional chemotherapy, large-area radiotherapy, immune therapy or any biological anti-tumor therapy 4 weeks before enrollment;
* allergic to ingredients in this trial;
* common terminology criteria for adverse events ≥2 because of the previous surgery or treatment-related adverse reactions;
* with two types of primary solid tumors;
* poorly managed hypertension (systolic blood pressure >160 mmHg and / or diastolic blood pressure > 90 mmHg) or clinically serious (for example, active) cerebrovascular diseases such as cerebrovascular incident (within 6 months prior to signing the informed consent), myocardial infarction (within 6 months prior to signing the informed consent), unstable angina, grade II or above heart failure according to New York Heart Association Grading Congestive, or severe arrhythmia can not be controlled by medication or has a potential impact on the study; with consecutive three times of obvious abnormality on electrocardiogram or average QT corrected interval ≥450 millisecond;
* combined with other serious organic and mental disorders;
* serious or active bacteria, viral or fungal infections that require systemic treatment;
* with autoimmune diseases: such as a history of inflammatory bowel disease or other autoimmune diseases determined by the investigator as unsuitable for the study (e.g. systemic lupus erythematosus,vasculitis, invasive pulmonary disease);
* within 4 weeks prior the infusion, received chronic systemic steroid cortisone, hydroxyurea, immunomodulatory treatment (for example: Interleukin 2, alpha or gamma interferon, granulocyte colony stimulating factor, mammalian target of rapamycin inhibitors, cyclosporine, Thymosin etc);
* with organ transplantation, autologous/allogeneic stem cell transplantation and renal replacement therapy;
* with central nervous system metastasis but not receive treatment;
* with uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease, or liver failure;
* alcohol and / or drug abuse;
* pregnant or lactating women;
* received concomitant medication prohibited by this trial;
* with any medical condition or disease determined by the investigators that may be detrimental to this trial;
* without legal capacity / limited behavior.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
treatment-related adverse events as assessed by CTCAE v4.03 | 28 Days
  The treatment-related adverse events of the patients received TAEST16001 treatment will be assessed by CTCAE v4.03

SECONDARY OUTCOMES:
assess overall response rate | 270 Days
  The overall response rate is evaluated according to Response Evaluation Criteria In Solid Tumors or Immune Related Response Criteria
assess duration of response | 270 Days
  The efficacy of TAEST16001 will be assessed by duration of response(DOR).The DOR refers to the length of time from the first appearance of a treatment response to the first occurrence of progressive disease or recurrence.
assess time to progress | 270 Days
  The efficacy of TAEST16001 will be assessed by time to progress (TTP).The TTP refers to the time from treatment to disease progression
assess progression free survival | 270 Days
  The efficacy of TAEST16001 will be assessed by progression free survival (PFS).The PFS refers to the time from treatment to progressive disease or death for any reason
assess overall survival | 270 Days
  The efficacy of TAEST16001 will be assessed by overall survival (OS).The OS refers to the time from treatment to death
assess the expression of tumor markers | 270 Days
  The efficacy of TAEST16001 will be assessed by tumor markers including carcinoembryonic antigen,carbohydrate antigen199,carbohydrate antigen125,prostate specific antigen,alpha fetoprotein,carbohydrate antigen724.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Study Chair — Southern Medical University, China
Locations (1):
- Zhujiang Hospital of Southern Mediacl University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rapoport AP, Stadtmauer EA, Binder-Scholl GK, Goloubeva O, Vogl DT, Lacey SF, Badros AZ, Garfall A, Weiss B, Finklestein J, Kulikovskaya I, Sinha SK, Kronsberg S, Gupta M, Bond S, Melchiori L, Brewer JE, Bennett AD, Gerry AB, Pumphrey NJ, Williams D, Tayton-Martin HK, Ribeiro L, Holdich T, Yanovich S, Hardy N, Yared J, Kerr N, Philip S, Westphal S, Siegel DL, Levine BL, Jakobsen BK, Kalos M, June CH. NY-ESO-1-specific TCR-engineered T cells mediate sustained antigen-specific antitumor effects in myeloma. Nat Med. 2015 Aug;21(8):914-921. doi: 10.1038/nm.3910. Epub 2015 Jul 20. PMID 26193344
- [Background] Li Y, Moysey R, Molloy PE, Vuidepot AL, Mahon T, Baston E, Dunn S, Liddy N, Jacob J, Jakobsen BK, Boulter JM. Directed evolution of human T-cell receptors with picomolar affinities by phage display. Nat Biotechnol. 2005 Mar;23(3):349-54. doi: 10.1038/nbt1070. Epub 2005 Feb 20. PMID 15723046
- [Background] Robbins PF, Kassim SH, Tran TL, Crystal JS, Morgan RA, Feldman SA, Yang JC, Dudley ME, Wunderlich JR, Sherry RM, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Li YF, El-Gamil M, Rosenberg SA. A pilot trial using lymphocytes genetically engineered with an NY-ESO-1-reactive T-cell receptor: long-term follow-up and correlates with response. Clin Cancer Res. 2015 Mar 1;21(5):1019-27. doi: 10.1158/1078-0432.CCR-14-2708. Epub 2014 Dec 23. PMID 25538264
- [Background] Robbins PF, Morgan RA, Feldman SA, Yang JC, Sherry RM, Dudley ME, Wunderlich JR, Nahvi AV, Helman LJ, Mackall CL, Kammula US, Hughes MS, Restifo NP, Raffeld M, Lee CC, Levy CL, Li YF, El-Gamil M, Schwarz SL, Laurencot C, Rosenberg SA. Tumor regression in patients with metastatic synovial cell sarcoma and melanoma using genetically engineered lymphocytes reactive with NY-ESO-1. J Clin Oncol. 2011 Mar 1;29(7):917-24. doi: 10.1200/JCO.2010.32.2537. Epub 2011 Jan 31. PMID 21282551
- [Background] Johnson LA, Morgan RA, Dudley ME, Cassard L, Yang JC, Hughes MS, Kammula US, Royal RE, Sherry RM, Wunderlich JR, Lee CC, Restifo NP, Schwarz SL, Cogdill AP, Bishop RJ, Kim H, Brewer CC, Rudy SF, VanWaes C, Davis JL, Mathur A, Ripley RT, Nathan DA, Laurencot CM, Rosenberg SA. Gene therapy with human and mouse T-cell receptors mediates cancer regression and targets normal tissues expressing cognate antigen. Blood. 2009 Jul 16;114(3):535-46. doi: 10.1182/blood-2009-03-211714. Epub 2009 May 18. PMID 19451549
- [Background] Morgan RA, Dudley ME, Wunderlich JR, Hughes MS, Yang JC, Sherry RM, Royal RE, Topalian SL, Kammula US, Restifo NP, Zheng Z, Nahvi A, de Vries CR, Rogers-Freezer LJ, Mavroukakis SA, Rosenberg SA. Cancer regression in patients after transfer of genetically engineered lymphocytes. Science. 2006 Oct 6;314(5796):126-9. doi: 10.1126/science.1129003. Epub 2006 Aug 31. PMID 16946036